CLINICAL TRIAL: NCT00001803
Title: Von Hippel-Lindau (VHL) Disease Genetic Epidemiology Study
Brief Title: Von Hippel-Lindau Disease Genetic Epidemiology Study
Status: Terminated | Type: Observational
Why Stopped: IRB approval lapsed and PI has not responded to requests to submit CR.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990053; 99-C-0053; NCT00003866 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Von Hippel Lindau Disease; Kidney Neoplasms
Keywords: Gene-Environment Interaction; Kidney Cancer; VHL; Genetic Epidemiology
MeSH Terms: conditions — von Hippel-Lindau Disease; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
The Von Hippel-Lindau (VHL) Disease Genetic Epidemiology Study is a family-based case-control study to be conducted by the National Cancer Institute. The study subjects are 603 individuals who were determined to belong to families with VHL disease confirmed through screening under NIH protocol #89-C-0086 between 1988 and 1998. There are 293 patient volunteers with VHL disease and 310 volunteer patients free of VHL disease, most of whom have already had genetic testing for mutations in the VHL gene. Adults as well as children aged 13 - 17 will be included. All subjects will give informed consent prior to participation; for minor subjects, assent will be obtained from the minor and consent from the parent/guardian. This protocol provides the potential to benefit people with VHL disease (although not necessarily the study subjects themselves) and possibly people with sporadic (non-hereditary) forms of the tumors which occur in VHL disease. The risks and discomfort associated with this study are minor.

The present protocol is a new epidemiologic component to VHL research at NIH which will relate the expression of VHL tumors to lifestyle factors (tobacco and alcohol use; physical activity), occupational exposures, reproductive and hormonal factors, demographic factors, medication use, diet, and putative susceptibility genes. Information will be collected by telephone interview and a written, self-administered diet questionnaire. A cheek cell sample will be obtained for analyses of genetic polymorphisms. Medical records will be obtained to document events reported by the subject at interview. Primary comparisons will be between VHL patients with a particular manifestation and VHL patients who are free of that condition. Additional comparisons may be made with unaffected family members who lack a mutation in the VHL gene, as appropriate.

DETAILED DESCRIPTION:
The Von Hippel-Lindau (VHL) Disease Genetic Epidemiology Study is a family-based case-control study to be conducted by the National Cancer Institute. The study subjects are 603 individuals who were determined to belong to families with VHL disease confirmed through screening under NIH protocol #89-C-0086 between 1988 and 1998. There are 293 patient volunteers with VHL disease and 310 volunteer patients free of VHL disease, most of whom have already had genetic testing for mutations in the VHL gene. Adults as well as children aged 13 - 17 will be included. All subjects will give informed consent prior to participation; for minor subjects, assent will be obtained from the minor and consent from the parent/guardian. This protocol provides the potential to benefit people with VHL disease (although not necessarily the study subjects themselves) and possibly people with sporadic (non-hereditary) forms of the tumors which occur in VHL disease. The risks and discomfort associated with this study are minor.

The present protocol is a new epidemiologic component to VHL research at NIH which will relate the expression of VHL tumors to lifestyle factors (tobacco and alcohol use; physical activity), occupational exposures, reproductive and hormonal factors, demographic factors, medication use, diet, and putative susceptibility genes. Information will be collected by telephone interview and a written, self-administered diet questionnaire. A cheek cell sample will be obtained for analyses of genetic polymorphisms. Medical records will be obtained to document events reported by the subject at interview. Primary comparisons will be between VHL patients with a particular manifestation and VHL patients who are free of that condition. Additional comparisons may be made with unaffected family members who lack a mutation in the VHL gene, as appropriate.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible patient volunteers are those who:

1. have been enrolled in protocol 89-C-0086;
2. are a member of a family in which at least one person has been diagnosed with VHL at NIH; and
3. are at least 13 years of age.

Patient volunteers seen under protocol 89-C-0086 who have been diagnosed with VHL, are at risk of VHL, or are unaffected are all eligible for study.

Additional families screened throughout the field period and meeting all eligibility criteria will also be able to participate.

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 1999-02-26; Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
To relate the expression of VHL tumors to lifestyle factors (tobacco & alcohol use, physical activity), occupational exposures, reproductive and hormonal factors, demographic factors, medication use, diet, and putative susceptibility gen... | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Neil E Caporaso, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chow WH, Gridley G, McLaughlin JK, Mandel JS, Wacholder S, Blot WJ, Niwa S, Fraumeni JF Jr. Protein intake and risk of renal cell cancer. J Natl Cancer Inst. 1994 Aug 3;86(15):1131-9. doi: 10.1093/jnci/86.15.1131. PMID 8028035
- [Background] Neumann HP, Zbar B. Renal cysts, renal cancer and von Hippel-Lindau disease. Kidney Int. 1997 Jan;51(1):16-26. doi: 10.1038/ki.1997.3. No abstract available. PMID 8995713
- [Background] Chen F, Kishida T, Yao M, Hustad T, Glavac D, Dean M, Gnarra JR, Orcutt ML, Duh FM, Glenn G, et al. Germline mutations in the von Hippel-Lindau disease tumor suppressor gene: correlations with phenotype. Hum Mutat. 1995;5(1):66-75. doi: 10.1002/humu.1380050109. PMID 7728151
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-C-0053.html